CLINICAL TRIAL: NCT01223950
Title: Monitoring the Prevalence of E.R Admissions and Hospitalizations as a Result of Drug Related Problems (DRPs)
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Jalal Ashkar MD, Eyal Schawartzberg, Hillel Yaffe medical center
Other Study IDs: 0067-10-HYMC
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Drug Related Problems Associated Hospitalizations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To research the prevalence and nature of DRP (Drug Related Problems) associated hospitalizations (hospitalizations due to problems\adverse effects of the medication treatment) .

Analyzing the main reasons for DRP associated E.R admissions\hospitalizations. identifying drug involved and percentage of DRP associated hospitalizations.

Monitoring the length of DRP associated hospitalizations. Evaluating LOS to hospitalized. Financial and other aspects will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Possible DRP based on the current literature, patient questionnaire and drug history, related laboratories test values, ICD-9 coding.

Exclusion Criteria:

* DRP cannot be established or suspected based on the assessment of the patient's lab results, symptoms, drug treatment and patient's questioning as well as physician diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age and above) admitted to the E.R and subsequently to hospital wards of the Hillel Yaffe medical center, Hadera, Israel.
Sampling Method: Non-Probability Sample
Enrollment: 12350 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual)

REFERENCES:
- [Background] Doggrell SA. Adherence to medicines in the older-aged with chronic conditions: does intervention by an allied health professional help? Drugs Aging. 2010 Mar 1;27(3):239-54. doi: 10.2165/11532870-000000000-00000. PMID 20210369
- [Background] Sotoca Momblona JM, Canivell Fuste S, Alemany Vilches L, Siso Almirall A, Codina Jane C, Ribas Sala J. [Drug related problems and hospital admissions]. Aten Primaria. 2009 Mar;41(3):141-6. doi: 10.1016/j.aprim.2008.07.002. Epub 2009 Apr 8. Spanish. PMID 19356826
- [Background] Rogers S, Wilson D, Wan S, Griffin M, Rai G, Farrell J. Medication-related admissions in older people: a cross-sectional, observational study. Drugs Aging. 2009;26(11):951-61. doi: 10.2165/11316750-000000000-00000. PMID 19848440
- [Background] Al-Olah YH, Al Thiab KM. Admissions through the emergency department due to drug-related problems. Ann Saudi Med. 2008 Nov-Dec;28(6):426-9. doi: 10.5144/0256-4947.2008.426. PMID 19011316
- [Background] Howard R, Avery A, Bissell P. Causes of preventable drug-related hospital admissions: a qualitative study. Qual Saf Health Care. 2008 Apr;17(2):109-16. doi: 10.1136/qshc.2007.022681. PMID 18385404
- [Background] Blix HS, Viktil KK, Moger TA, Reikvam A. Characteristics of drug-related problems discussed by hospital pharmacists in multidisciplinary teams. Pharm World Sci. 2006 Jun;28(3):152-8. doi: 10.1007/s11096-006-9020-z. Epub 2006 Sep 27. PMID 17004023
- [Background] Koh Y, Fatimah BM, Li SC. Therapy related hospital admission in patients on polypharmacy in Singapore: a pilot study. Pharm World Sci. 2003 Aug;25(4):135-7. doi: 10.1023/a:1024896328720. PMID 12964490
- [Background] Patel P, Zed PJ. Drug-related visits to the emergency department: how big is the problem? Pharmacotherapy. 2002 Jul;22(7):915-23. doi: 10.1592/phco.22.11.915.33630. PMID 12126224
- [Background] Klein C, Prokhorov T, Miniovitz A, Dobronevsky E, Rabey JM. Admission of Parkinsonian patients to a neurological ward in a community hospital. J Neural Transm (Vienna). 2009 Nov;116(11):1509-12. doi: 10.1007/s00702-009-0302-1. PMID 19763774